CLINICAL TRIAL: NCT00294775
Title: Left Ventricular Reverse Remodelling After Aortic Valve Replacement in Severe Valvular Aortic Stenosis - Effect of Blockade of the Angiotensin-II Receptor
Brief Title: Effect of Angiotensin II Receptor Blockers (ARB) on Left Ventricular Reverse Remodelling After Aortic Valve Replacement in Severe Valvular Aortic Stenosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT number 2005-001930-34
Record Dates: First submitted 2006-02-21; First posted 2006-02-22 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Aortic Valve Stenosis; Left Ventricular Hypertrophy; Atrial Fibrillation
Keywords: diastolic dysfunction; Reverse Remodelling
MeSH Terms: conditions — Aortic Valve Stenosis; Hypertrophy, Left Ventricular; Atrial Fibrillation | interventions — candesartan

INTERVENTIONS:
Drug: Candesartan

SUMMARY:
The consequence of aortic valve stenosis (AVS) is increased pressure load on the left ventricle which causes left ventricular (LV) hypertrophy, and myocardial stretch will cause activation of cardiac peptides and activation of the renin angiotensin aldosterone system (RAAS). The consequence of LV hypertrophy is increased chamber-stiffness and delayed active LV relaxation which initially will cause diastolic and later systolic dysfunction. In heart failure (HF) and ischemic heart disease the degree of diastolic dysfunction has been demonstrated to correlate with functional class, neurohormonal activation and prognosis which also recently have been suggested for AVS.

With longstanding elevated filling pressures the left atrium (LA) will dilate. Only limited data are available on the degree and importance of LA dilatation in AVS.

When apparent, symptoms of HF in AVS are associated with high mortality rates. If LV systolic dysfunction also is present prognosis will deteriorate further. In these cases aorta valve replacement (AVR) is recommended. AVR will normalize pressure overload and thereby decreases LV hypertrophy. Previously it was believed that in time LV hypertrophy regressed towards normal and even normalized. Recent studies however have demonstrated that LV hypertrophy regression mainly happens during the first year after AVR, and little subsequent changes are seen during the remaining 10 years. Furthermore, patients that experience most regression of hypertrophy have more favourable outcome and better functional class than patients with less regression of hypertrophy. Thus absence of reverse remodelling is associated with poor outcome after AVR. Importantly the regression of LV hypertrophy is closely paralleled by decreasing RAAS hyperactivity.

RAAS hyperactivity may be attenuated pharmacologically with angiotensin II receptor blockers (ARB) which in systemic hypertension with LV hypertrophy has been associated with reverse remodelling.

The hypothesis is that in patients undergoing AVR for symptomatic AVS, 12 months post operative blockade of the angiotensin II receptor will accelerate LV and LA reverse remodelling, reduce filling pressures and suppress neurohormonal activation compared with conventional therapy. This will lead to improved exercise tolerance and due to improved left atrial function reducing the risk of atrial arrythmias.

DETAILED DESCRIPTION:
1. Background:

   Aortic valve stenosis (AVS) is the most common valvular disease in the western world. The prevalence increases with age where "degenerative" changes of the aortic valve with thickening, accumulation of calcium and progressive dysfunction of the valve usually becomes apparent in patients older than 60 years. Although the development of AVS generally is believed to be a degenerative process more recent studies have demonstrated AVS is caused by a complex process of increased cellularity, lipid accumulation, extracellular matrix deposition, and with disease progression calcification of lesions. Although mild and moderate AVS generally is well tolerated severe AVS is associated with considerable morbidity and mortality, and valve replacement is generally required.

   The consequence of AVS is increased pressure load on the left ventricle which causes changes in the ventricular structure. Pressure overload causes replication of the sarcomeres leading to left ventricular (LV) hypertrophy, and myocardial stretch will cause activation of cardiac peptides and activation of the renin angiotensin aldosterone system (RAAS). With progression of disease, RAAS activation will, through stimulation of the angiotensin-II receptor mediate fibroblast proliferation, promote fibrosis and directly affect the extracellular matrix. The consequence of LV hypertrophy and interstitial fibrosis is increased chamber-stiffness and delayed active LV relaxation which initially will cause diastolic (increased LV end-diastolic pressure) and later in the disease progression also systolic dysfunction. In congestive heart failure and ischemic heart disease the degree of diastolic dysfunction has been demonstrated to correlate with functional class, neurohormonal activation and prognosis which also recently has been suggested for AVS. Thus, although not fully elucidated the transition from well compensated hypertrophy caused by pressure overload to symptomatic heart failure may be related to evolving diastolic dysfunction. With longstanding elevated filling pressures the left atrium will dilate due to chronically increased atrial afterload. Only limited data are available on the degree and importance of LA dilatation in AVS.

   When apparent, symptoms of heart failure in AVS is associated with high mortality rates. If LV systolic dysfunction also is present prognosis will deteriorate further. In these cases aorta valve replacement (AVR) is recommended. AVR will normalize pressure overload and thereby decreases LV hypertrophy. Previously it was believed that in time LV hypertrophy regressed towards normal and even normalized. More recent studies however have demonstrated that LV hypertrophy regression mainly happens during the first 12-18 months after AVR, and little subsequent changes are seen during the remaining 10 years. Furthermore, patients that experience most regression of hypertrophy has more favourable outcome and better functional class than patients with less regression of hypertrophy. Thus absence of reverse remodelling is associated with poor outcome after AVR. Importantly the regression of LV hypertrophy is closely paralleled by decreasing RAAS hyperactivity.

   RAAS hyperactivity may be attenuated pharmacologically using angiotensin converting enzyme inhibitors (ACEi) or angiotensin II receptor blockers (ARB) which in systemic hypertension with LV hypertrophy has been associated with reverse remodelling. This may at least partly be associated with increased collagenase activity and depressed collagen synthesis. Thus attenuation of RAAS hyperactivity may in theory lead to decreased myocardial fibrosis and improving the diastolic function of the LV. The effect of ARB treatment in patients with AVS that have undergone AVR is not known.
2. Hypothesis:

   In patients undergoing AVR for symptomatic valvular aortic stenosis, 12 months post operative blockade of the angiotensin II receptor will accelerate LV and LA reverse remodelling, reduce filling pressures and suppress neurohormonal activation compared with conventional therapy. This will lead to improved exercise tolerance and due to improved left atrial function reducing the risk of atrial arrythmias.
3. Specific Objectives:

   3.1 Primary Objectives
   * In a consecutive population undergoing AVR for symptomatic AVS to compare

     1. LV mass index
     2. LA volume index
     3. Plasma nt-pro BNP concentration after 12 months treatment with candesartan compared with conventional treatment

   3.2 Secondary Objectives
   * In a consecutive population undergoing AVR for symptomatic AVS to compare

     1. Diastolic E/e' ratio
     2. Overall LV function assessed by the Doppler echocardiographic Tei Index
     3. Regional LV function assessed with tissue Doppler imaging
     4. LV end systolic and end diastolic volume index after 12 months treatment with candesartan compared with conventional treatment.

   3.3 Tertiary Objectives
   * In a consecutive population undergoing AVR for symptomatic AVS to compare the occurrence and atrial arrhythmias assessed with 48h Holter after 12 months treatment with candesartan compared with conventional management.
   * In a consecutive population undergoing AVR for symptomatic AVS to compare exercise capacity after 12 months treatment with candesartan compared with conventional management.
   * In a consecutive population undergoing AVR for symptomatic AVS to assess serial changes in LV diastolic, overall LV function and regional LV systolic function 12 months after valve replacement
   * In a consecutive population undergoing AVR for symptomatic AVS to assess serial changes in plasma nt-pro BNP, ANP, and renin 12 months after valve replacement.
4. Methods:

4.1 Design

The study is a prospective single center randomized study (PROBE design). Eligible patients will be randomized to either conventional management or conventional management and 12 months treatment with candesartan. Treatment with candesartan will be unblinded but all neurohormonal analyses and analyses of LV and LA size and function will be performed blinded for treatment allocation and clinical data.

4.4 Study Procedures

Patients scheduled for elective aortic valve replacement for severe AVS at Odense University Hospital will consecutively be offered participation in the study at hospital admission (2 days prior to surgery). If patient consent is obtained patients will undergo the study program. Baseline echocardiography, neurohormonal analyses, and 6 min walk test will be performed the day before surgery. After surgery and when the patient is transferred from cardiac intensive care unit to step down unit treatment with candesartan (Atacand®) 8 mg daily is initiated, and during hospitalization patients are titrated to 32 mg. After hospital discharge patients will be followed in the heart failure clinic at Odense University Hospital. Study medication will be handed to the patient at each visit.

Enrollment is planned to start February 2006 and continue for 18 months or until 140 patients have been enrolled.

4.4.1 Echocardiography

Doppler echocardiography will be performed prior to valve replacement, and repeated 3, 6, and 12 months after surgery. Examinations will be performed on a GE medical Vivid 5 ultrasound machine. Images will be obtained from the parasternal and apical windows. M-mode recordings will be done in the parasternal long-axis view. Pulsed Doppler measurements of mitral inflow will be obtained with the transducer in the apical four-chamber view, with a 1-2 mm Doppler sample volume placed between the tips of mitral leaflets during diastole. Tissue Doppler imaging of the mitral annulus will be obtained from the apical 4-chamber view with a 1.5-mm sample volume placed at the medial mitral annulus. All Doppler echocardiographic examinations are done with horizontal sweep set to 100 mm/s. At least 3-5 cardiac cycles will be measured. Finally color coded real time tissue Doppler images will be acquired in the apical windows.

* End-systolic, end-diastolic volume and ejection fraction will be calculated according to the Simpson modified biplane method.
* LV mass will be estimated using the recommendations of the American Society of Echocardiography.
* Maximal left atrial volume will be measured at end-systole with the use of two orthogonal apical views.
* From the pulsed wave mitral inflow signal, peak E wave velocity, peak A wave velocity, and mitral E-wave deceleration time will be measured. From pulsed wave Doppler recording of LV outflow ejection time will be recorded. From these recordings Tei index will be assessed.
* From peak tricuspid regurgitant velocity and size of inferior v. cava pulmonary arterial systolic pressure will be estimated.
* From the tissue Doppler assessment of the medial mitral annulus early (E') diastolic velocity will be recorded. Diastolic function will be graded in grades 0-3 and diastolic E/e' ratio calculated.
* From color coded tissue Doppler images systolic longitudinal fibre shortening will be assessed using tissue tracking, and systolic strain will be assessed on a regional basis.

4.4.2 Neurohormonal Analyses

Prior to surgery and at each follow-up visit venous blood samples will be drawn for analysis of plasma N-terminal proBNP, and of plasma N-terminal ANP concentrations. In addition prior to surgery and after 6 and 12 months treatment with candesartan RAAS activity will be assessed using plasma-renin activity, plasma-aldosterone, and plasma-noradrenalin. In addition plasma will be frozen at each visit for possible later analysis.

4.4.3 Six Minutes Walk Test

A 6 min. walk test will be performed at baseline and at each outpatient visit (3, 6, 9 and 12 month).

4.4.3 Holter Monitoring

At the 12 months visit a 2-channel 48 hours Holter monitoring will be performed and analyzed for occurrence of atrial arrhythmias.

4.4.4 Blood Pressure

Measurement of blood pressure will be done standardized after 30 min of rest at each visit. Target blood pressure will be 140/80 mmHg or less and treatment instituted when appropriate.

4.4.5 Study Events

During the study period hospitalizations for worsening of heart failure, fatal / nonfatal stroke, fatal/nonfatal acute coronary syndrome, hospitalization for atrial arrhythmias, and death from all causes will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic severe AVS referred for valve replacement (mechanic prosthesis or bioprosthesis) at Odense University Hospital
2. Signed informed consent

Exclusion Criteria:

1. Severe renal failure (s-creatinine >300 mmole/l)
2. Moderate or severe hepatic failure
3. Moderate or severe LV systolic dysfunction (LVEF<40%)
4. Patients already treated with ACE-I or ARB
5. Known intolerance for ARB
6. Unwilling to participate in the study
7. Poor echocardiographic window
8. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2006-02; Primary Completion 2009-01 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
LV mass index
LA volume index
Plasma nt-pro BNP concentration

SECONDARY OUTCOMES:
Diastolic E/e' ratio
Overall LV function assessed by the Doppler echocardiographic Tei Index
Regional LV function assessed with tissue Doppler imaging
LV end systolic and end diastolic volume index
Atrial arrhythmias assessed with 48h Holter after 12 months
Exercise capacity after 12 months
Serial changes in LV diastolic, overall LV function and regional LV systolic function
Assess serial changes in plasma nt-pro BNP, ANP, and renin

CONTACTS AND LOCATIONS:
Overall Officials: Torben Haghfelt, Md, DMSc, Study Director — Kardiologisk forskningsenhed, OUH; Jordi S Dahl, MD, MMSci, Principal Investigator — Kardiologisk forskningsenhed, OUH; Henrik Nissen, MD, PhD, Study Chair — Kardiologisk forskningsenhed, OUH; Jacob E Moller, Md, Ph.D, Study Chair — Kardiologisk forskningsenhed, OUH; Lars Videbæk, MD, Ph.d, Study Chair — Kardiologisk forskningsenhed, OUH; Lars I Andersen, MD, DMSc, Study Chair — Department of thoracic surgery, OUH
Locations (1):
- Cardiology Department, Odense University hospital, Odense, Fyn, Denmark

REFERENCES:
- [Background] Lindroos M, Kupari M, Heikkila J, Tilvis R. Prevalence of aortic valve abnormalities in the elderly: an echocardiographic study of a random population sample. J Am Coll Cardiol. 1993 Apr;21(5):1220-5. doi: 10.1016/0735-1097(93)90249-z. PMID 8459080
- [Background] Walther T, Schubert A, Falk V, Binner C, Walther C, Doll N, Fabricius A, Dhein S, Gummert J, Mohr FW. Left ventricular reverse remodeling after surgical therapy for aortic stenosis: correlation to Renin-Angiotensin system gene expression. Circulation. 2002 Sep 24;106(12 Suppl 1):I23-6. PMID 12354704
- [Background] Walther T, Schubert A, Falk V, Binner C, Kanev A, Bleiziffer S, Walther C, Doll N, Autschbach R, Mohr FW. Regression of left ventricular hypertrophy after surgical therapy for aortic stenosis is associated with changes in extracellular matrix gene expression. Circulation. 2001 Sep 18;104(12 Suppl 1):I54-8. doi: 10.1161/hc37t1.094777. PMID 11568030
- [Background] Giorgi D, Di Bello V, Talini E, Palagi C, Delle Donne MG, Nardi C, Verunelli F, Mariani MA, Di Cori A, Caravelli P, Mariani M. Myocardial function in severe aortic stenosis before and after aortic valve replacement: a Doppler tissue imaging study. J Am Soc Echocardiogr. 2005 Jan;18(1):8-14. doi: 10.1016/j.echo.2004.08.012. PMID 15637482
- [Background] Lund O, Emmertsen K, Dorup I, Jensen FT, Flo C. Regression of left ventricular hypertrophy during 10 years after valve replacement for aortic stenosis is related to the preoperative risk profile. Eur Heart J. 2003 Aug;24(15):1437-46. doi: 10.1016/s0195-668x(03)00316-6. PMID 12909073
- [Derived] Sabino-Carvalho JL, Li S, Mekonnen E, Mammino K, Nocera JR, Park J. Aerobic Cycling Exercise Training Does Not Improve Impaired Vagal Reactivation in Patients with Chronic Kidney Disease. Med Sci Sports Exerc. 2025 Dec 1;57(12):2621-2629. doi: 10.1249/MSS.0000000000003824. Epub 2025 Jul 16. PMID 40665514
- [Derived] Dahl JS, Barros-Gomes S, Videbaek L, Poulsen MK, Issa IF, Carter-Storch R, Christensen NL, Kumme A, Pellikka PA, Moller JE. Early Diastolic Strain Rate in Relation to Systolic and Diastolic Function and Prognosis in Aortic Stenosis. JACC Cardiovasc Imaging. 2016 May;9(5):519-28. doi: 10.1016/j.jcmg.2015.06.029. Epub 2016 Apr 13. PMID 27085434
- [Derived] Dahl JS, Christensen NL, Videbaek L, Poulsen MK, Carter-Storch R, Hey TM, Pellikka PA, Steffensen FH, Moller JE. Left ventricular diastolic function is associated with symptom status in severe aortic valve stenosis. Circ Cardiovasc Imaging. 2014 Jan;7(1):142-8. doi: 10.1161/CIRCIMAGING.113.000636. Epub 2013 Oct 30. PMID 24173271
- [Derived] Dahl JS, Moller JE, Videbaek L, Poulsen MK, Rudbaek TR, Pellikka PA, Scott Argraves W, Rasmussen LM. Plasma fibulin-1 is linked to restrictive filling of the left ventricle and to mortality in patients with aortic valve stenosis. J Am Heart Assoc. 2012 Dec;1(6):e003889. doi: 10.1161/JAHA.112.003889. Epub 2012 Dec 19. PMID 23316326
- [Derived] Dahl JS, Videbaek L, Poulsen MK, Rudbaek TR, Pellikka PA, Moller JE. Global strain in severe aortic valve stenosis: relation to clinical outcome after aortic valve replacement. Circ Cardiovasc Imaging. 2012 Sep 1;5(5):613-20. doi: 10.1161/CIRCIMAGING.112.973834. Epub 2012 Aug 6. PMID 22869821
- [Derived] Dahl JS, Videbaek L, Poulsen MK, Pellikka PA, Veien K, Andersen LI, Haghfelt T, Moller JE. Noninvasive assessment of filling pressure and left atrial pressure overload in severe aortic valve stenosis: relation to ventricular remodeling and clinical outcome after aortic valve replacement. J Thorac Cardiovasc Surg. 2011 Sep;142(3):e77-83. doi: 10.1016/j.jtcvs.2011.01.032. Epub 2011 Feb 25. PMID 21353251